CLINICAL TRIAL: NCT02886351
Title: High-Concentration Nitrous Oxide for Dental Procedural Sedation in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, MOSTAFA.SOMRI, M.D., Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BnaiZionMC-16-MS-002
Record Dates: First submitted 2016-08-28; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Anxiety
Keywords: Moderate Sedation; Pediatric Dentistry; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Nitrous Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nitrous oxide (Experimental): Administration of high concentration of nitrous oxygen in pediatric dentistry
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous Oxide at 60%-70% concentration administrated by mask, to achieve cooperation in Pediatric dentisry
  Other Names: Dinitrogen monoxide; laugh gas

SUMMARY:
The use of nitrous oxide as a sedative agent is very common in pediatric dentistry. In concentrations up to 50% it is considered as mild sedation and it is very safe. Despite its safety and widespread of its use nitrous oxide is not a potent drug and many times dentists fail to gain cooperation in moderate or high anxious children, and the alternatives are to use moderate sedation with drugs such as Midazolam, Atarax or general anesthesia. Higher concentration was not conducted in Pediatry densitery. The aim of this study is to compare the effectivity and safety of providing nitrous oxide at increasing concentrations 60%, 70% with 50% parameters, sedation depth, adverse events and cooperation of the child during the dental treatment.Our hypothesis is that nitrous oxide in concentrations higher than 50% up to 70% is a safe and effective sedation method in dental treatment of children.

DETAILED DESCRIPTION:
Nitrous oxide/oxygen in varying concentrations has been successfully used for many years to provide sedation and analgesia for a variety of painful procedures in children. The use of nitrous oxide as a sedative agent is very common in pediatric dentistry. In concentrations up to 50% it is considered as mild sedation and it is very safe. It is usually used for mild or moderate anxiety state because it is not so potent in concentrations up to 50 %. Despite its safety and widespread of its use nitrous oxide is not a potent drug and many times dentists fail to gain cooperation in moderate or high anxious children, and the alternatives are to use moderate sedation with drugs such as Midazolam, Atarax or general anesthesia. Nitrous oxide 50% is the most common concentration in use but the results of the sedation does not always provide a satisfactory cooperation, higher concentration was not conducted in Pediatry densitery. The aim of this study is to compare the effectivity and safety of providing nitrous oxide at increasing concentrations 60%, 70% with 50% parameters, sedation depth, adverse events and cooperation of the child during the dental treatment.Our hypothesis is that nitrous oxide in concentrations higher than 50% up to 70% is a safe and effective sedation method in dental treatment of children.

ELIGIBILITY:
Inclusion Criteria:

* Children evaluated by a senior pediatric dentist and require a wide treatment of caries, with a high score of anxiety unable to accept dental treatment with nitrous oxide /oxide of 50% in combined with behavioral management in the pediatric dental clinic.

Exclusion criteria:

* Children with high potential risk of sedation, snoring, stridor, sleep apnea, maxillofacial malformation, history of airway difficulty, gastro esophageal reflux, reactive airway disease or acute runny nose, cardiac disease, altered mental status, inadequate fasting time.
* Parental refusal for conscious sedation.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Achieving cooperation in Pediatric dentistry numerical scale | less than 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Somri, M.D., Principal Investigator — Bnai Zion Medical Center

IPD SHARING:
Plan to Share IPD: Yes